CLINICAL TRIAL: NCT00991107
Title: A Phase I, Open Label Study of the Safety, Tolerance and Assessment of HE3286 on Insulin Sensitivity and Hepatic Glucose Production When Administered Orally to Obese Insulin-Resistant Adult Subjects for 28 Days
Brief Title: A Study of the Safety, Tolerance and Assessment of HE3286 on Insulin Sensitivity and Hepatic Glucose Production
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Harbor Therapeutics (Industry)
Responsible Party: Dwight R. Stickney, MD - Chief Medical Officer, Hollis-Eden Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE3286-0103
Record Dates: First submitted 2009-10-05; First posted 2009-10-07 (Estimated); Last update posted 2011-03-09 (Estimated); Status verified 2011-03

CONDITIONS: Insulin Resistance
Keywords: phase I; safety; tolerance; insulin resistance; obese
MeSH Terms: conditions — Insulin Resistance; Obesity | interventions — 17-ethynyl-5-androstene-3, 7, 17-triol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HE3286 (Experimental): HE3286 20 mg (10 mg BID)
  Interventions: Drug: HE3286

INTERVENTIONS:
Drug: HE3286 — HE3286 20 mg (10 mg BID) for 28 days
  Other Names: TRIOLEX

SUMMARY:
The objectives of this study are to evaluate the safety and tolerance of 20 mg (10 mg BID) of HE3286 when administered orally over 28 days to obese insulin-resistant adult subjects and, to assess the activity of HE3286 on insulin sensitivity and hepatic glucose production in obese insulin-resistant adult subjects.

DETAILED DESCRIPTION:
Hollis-Eden Pharmaceuticals, Inc. is developing a new class of therapeutics for the treatment of Type 2 diabetes mellitus (T2DM). The investigational drug, HE3286, is a synthetic analog of a naturally occurring hormone with a potentially new mechanism of action that may improve the current therapeutic options available to a T2DM patient.

The glucose clamp is the gold standard for measurement of insulin sensitivity. Given the observed activity of HE3286 in reducing insulin resistance in both impaired glucose intolerant subjects and type 2 diabetic patients, it is necessary to evaluate the physiological site of action (i.e. liver vs. skeletal muscle) of HE3286 in order to further understand the mechanism of action and to design future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject 18-65 years of age
* Body Mass Index (BMI) is at least 29 kg/m2 but no more than 35 kg/m2 for females and no more than 37 kg/m2 for males
* Subject has fasting blood glucose level of < 126 mg/dL at Screening
* Subject has a 2 hour postprandial (following 75 grams glucose administration) blood glucose of 140-200 mg/dL at Screening
* Subject has fasting plasma insulin >=10 μU/mL

Exclusion Criteria:

* Subject has a history of clinically significant cardiovascular disease (including coronary artery disease), clinically significant hepatic, respiratory or renal abnormalities, clinically significant endocrine disorders (including history of diabetes); or clinically significant neurological or psychiatric condition;
* Subject has any clinically significant abnormalities in laboratory results at screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerance of 20 mg (10 mg BID) of HE3286 when administered orally over 28 days to obese insulin-resistant adult subjects | Study duration and 1-month follow-up

SECONDARY OUTCOMES:
Activity of HE3286 on insulin sensitivity and hepatic glucose production in obese insulin-resistant adult subjects. | Study period (28-days)

CONTACTS AND LOCATIONS:
Overall Officials: Dwight R. Stickney, MD, Study Director — Harbor Therapeutics
Locations (1):
- Clinical Site, Baton Rouge, Louisiana, United States